CLINICAL TRIAL: NCT04670588
Title: A Prospective Observational Study to Determine the Feasibility of Tumor Response Assessment by Circulating Tumor DNA in Patients With Locally Advanced Rectal Cancer Undergoing Total Neoadjuvant Therapy
Brief Title: Response Assessment by Circulating Tumor DNA in Patients With Locally Advanced Rectal Cancer
Status: Withdrawn | Type: Observational
Why Stopped: No accrual.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sakti Chakrabarti, MD, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO00039395
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Rectal Cancer
Keywords: Locally advanced rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After obtaining informed consent, a venous blood sample and the archival tissue block from the initial diagnostic rectal tumor biopsy will be sent to the Natera laboratory for designing patient-specific ctDNA assay, which will be used to measure ctDNA levels in the peripheral venous blood samples at various time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Locally advanced rectal cancer patients: Patients with LARC undergoing TNT.
  Interventions: Diagnostic Test: Circulating tumor DNA(ctDNA) level measurement

INTERVENTIONS:
Diagnostic Test: Circulating tumor DNA(ctDNA) level measurement — The ctDNA level will be measured using the Signatera platform developed by Natera, Inc. Signatera is a patient-specific, tumor informed custom-built ctDNA monitoring assay.

SUMMARY:
This is a single-arm observational study to determine the feasibility of assessing tumor response utilizing Circulating tumor DNA (ctDNA) in patients of with locally advanced rectal cancer (LARC) undergoing standard-of-care total neoadjuvant therapy (TNT) consisting of systemic chemotherapy (modified FOLFOX or modified FOLFIRINOX) followed by concurrent chemoradiation (50.4 Gy over approximately six weeks with concurrent radiosensitizing dose of capecitabine/5-fluorouracil).

DETAILED DESCRIPTION:
In this observational study, patients with LARC who are selected for the standard-of-care TNT will be enrolled. After obtaining informed consent, a venous blood sample and the archival tissue block from the initial diagnostic rectal tumor biopsy will be sent to the Natera laboratory for designing patient-specific ctDNA assay, which will be used to measure ctDNA levels in the peripheral venous blood samples at various time points coinciding with the standard studies to assess tumor response. The blood sample needed for designing the assay and measuring the baseline ctDNA level will be obtained within four weeks before neoadjuvant chemotherapy begins. Subsequently, for patients undergoing 16 weeks of neoadjuvant chemotherapy, blood samples will be obtained for ctDNA level measurement at three time points ( after eight weeks/4 cycles of neoadjuvant chemotherapy within +/- 5 days of the magnetic resonance imaging (MRI) study, after 16 weeks/8 cycles of neoadjuvant chemotherapy within +/- 5 days of the MRI study, and one to 14 days before surgery ). For patients who receive eight weeks of neoadjuvant chemotherapy, two blood samples will be obtained for subsequent ctDNA measurements (after eight weeks/4 cycles of neoadjuvant chemotherapy within +/- 5 days of the MRI study, and one to 14 days before surgery). All patients may also choose to undergo additional serial ctDNA level measurements for surveillance after the surgery every three to four months for two years (optional).

Tumor response rate assessed by ctDNA (defined as reduction of ctDNA level at least by 90% compared to the baseline level) will be compared with the response rate assessed by the standard method (proctoscopic examination, pelvic MRI, etc.) to explore if a significant correlation exists between these two response assessment methods. If preliminary data support the hypothesis that peripheral blood ctDNA can be utilized for tumor response assessment in this scenario, a larger study will be conducted to validate this method. Once validated, ctDNA measurement can potentially replace expensive, uncomfortable, and time-consuming methods of tumor response assessment like MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically documented rectal cancer eligible for total neoadjuvant therapy (TNT).
2. Male or female subjects ≥18 years old.
3. Rectal tumor biopsy is available for SignateraTM assay development for ctDNA measurement.
4. Patients must be able to understand the informed consent form and provide written consent.

Exclusion Criteria:

1. Patients without available rectal biopsy tissue for SignateraTM assay development.
2. Patients with rectal cancer not eligible to receive standard-of-care TNT for any reason.
3. Patients with undetectable ctDNA level in the baseline blood sample.
4. Patients without trackable mutation in the rectal tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer (LARC) undergoing total neoadjuvant therapy (TNT).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Mean serum ctDNA concentration | Baseline, 8 weeks, 16 weeks, around 24 weeks before rectal surgery.
  This measure is the concentration of ctDNA in plasma expressed as mean tumor molecules (MTM)/ml at specific time points.

SECONDARY OUTCOMES:
Response based on serum ctDNA level (change from baseline) | Baseline, 8 weeks, 16 weeks, around 24 weeks before rectal surgery
  This measure is the number of subjects achieving a reduction of ctDNA level (mean tumor molecules[MTM]/ml) by > 90% compared to the baseline.
Response based on standard clinical assessments | Baseline, 8 weeks, 16 weeks, around 24 weeks before rectal surgery.]
  This measure is the number of subjects achieving a clinical change of tumor size based on standard clinical assessments. Response will be a determined as a subjective measure by experienced clinicians using any combination of pelvic MRI, visual proctoscopic examination, sigmoidoscopy, and/or endoscopic ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Sakti Chakrabarti, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- See also: Manufacturer's site posting four scientific abstracts. — https://www.natera.com/oncology/signatera-clinicians